CLINICAL TRIAL: NCT04895878
Title: Patients With Co-occurrence of ANCA Vasculitis and Sjögren Syndrome : a Case Series and Systematic Review
Brief Title: Patients With Co-occurrence of ANCA Vasculitis and Sjögren Syndrome
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0288
Record Dates: First submitted 2021-05-10; First posted 2021-05-20 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: ANCA Associated Vasculitis; Sjogren's Syndrome
Keywords: Overlap syndrom
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ANCA vasculitis and Sjögren syndrome are two rare diseases, and even more rarely associated. These two conditions have specific organ involvements, and specific follow-up.

The Investigators hypothesise that patients with co-occurrence of these two diseases may have a singular clinical course.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of ANCA vasculitis based on clinical, immunological and histopathological features.
* Diagnosis of Sjögren syndrom based on ACR/EULAR 2016 criteria.

Exclusion criteria:

* Age < 18 years
* Insuffisant data during follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated in internal medicine services in secondary care centers of Languedoc-Roussillon region.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Severity of Sjögren disease | day 1 (Upon diagnosis)
  Severity of Sjögren disease

SECONDARY OUTCOMES:
Sjögren extra-glandular complications | day 1 (Upon diagnosis)
  Sjögren extra-glandular complications
severity of ANCA vasculitis | day 1 (Upon diagnosis)
  severity of ANCA vasculitis

CONTACTS AND LOCATIONS:
Overall Officials: Philippe GUILPAIN, MD, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Result] Guellec D, Cornec-Le Gall E, Groh M, Hachulla E, Karras A, Charles P, Dunogue B, Abad S, Alvarez F, Gerard F, Devauchelle-Pensec V, Pers JO, Puechal X, Guillevin L, Saraux A, Cornec D; CRI (Club Rhumatismes et Inflammation) and the French Vasculitis Study Group. ANCA-associated vasculitis in patients with primary Sjogren's syndrome: detailed analysis of 7 new cases and systematic literature review. Autoimmun Rev. 2015 Aug;14(8):742-50. doi: 10.1016/j.autrev.2015.04.009. Epub 2015 Apr 24. PMID 25916811
- [Result] Lee SB, Choi H, Kim MK, Jung SM, Song JJ, Park YB, Lee SW. Can antineutrophil cytoplasmic antibody positivity at diagnosis predict the poor outcomes of Sjogren's syndrome? Rheumatol Int. 2020 Jul;40(7):1063-1070. doi: 10.1007/s00296-019-04476-5. Epub 2019 Nov 12. PMID 31720749
- [Result] Ramos-Casals M, Brito-Zeron P, Font J. The overlap of Sjogren's syndrome with other systemic autoimmune diseases. Semin Arthritis Rheum. 2007 Feb;36(4):246-55. doi: 10.1016/j.semarthrit.2006.08.007. Epub 2006 Sep 22. PMID 16996579